CLINICAL TRIAL: NCT02856880
Title: A Study to Investigate the Antimicrobial Activity of Two Test Toothpastes in a Plaque Glycolysis and Regrowth Model
Brief Title: A Study to Investigate the Antimicrobial Activity of 2 Test Toothpastes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 205051
Record Dates: First submitted 2016-06-06; First posted 2016-08-05 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-07

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (5):
- Test zinc-IPMP toothpaste (Experimental): Rinse with preprepared slurry of toothpaste in 10 milliliter (mL) water for 60 seconds(s) followed by rinse with 10mL water
  Interventions: Other: Test zinc-IPMP toothpaste
- Test zinc non- IPMP toothpaste (Experimental): Rinse with preprepared slurry of toothpaste in 10 mL water for 60s followed by rinse with 10mL water
  Interventions: Other: Test zinc non- IPMP toothpaste
- Positive control Toothpaste (Active Comparator): Rinse with preprepared slurry of toothpaste in 10 mL water for 60s followed by rinse with 10mL water
  Interventions: Other: Positive control
- SLS Negative Control (Active Comparator): Rinse with preprepared slurry of toothpaste in 10 mL water for 60s followed by rinse with 10mL water
  Interventions: Other: SLS negative control
- non-SLS negative control (Active Comparator): Rinse with preprepared slurry of toothpaste in 10 mL water for 60s followed by rinse with 10mL water
  Interventions: Other: non-SLS negative control

INTERVENTIONS:
Other: Test zinc-IPMP toothpaste — Test toothpaste containing 0.6% w/w zinc chloride and 0.1% w/w IPMP and 1426ppm fluoride as sodium fluoride.
  Arms: Test zinc-IPMP toothpaste
Other: Test zinc non- IPMP toothpaste — Test toothpaste containing 0.6% w/w zinc chloride, 0% w/w IPMP and 1426ppm fluoride as sodium fluoride.
  Arms: Test zinc non- IPMP toothpaste
Other: Positive control — Positive control toothpaste containing 0.454% w/w stannous fluoride (Fluoride Toothpaste (1100ppm Fluoride as stannous fluoride)).
  Arms: Positive control Toothpaste
Other: SLS negative control — Negative control toothpaste containing 2.0% SLS, 0.65% Tegobetain and 1150 ppm fluoride as sodium fluoride
  Arms: SLS Negative Control
Other: non-SLS negative control — Negative control toothpaste containing 1426 ppm fluoride as sodium fluoride
  Arms: non-SLS negative control

SUMMARY:
The aim of this exploratory study is to assess the ability of two test toothpastes containing 0.6% w/w zinc chloride stabilised with sodium citrate in a sodium lauryl sulfate (SLS)-containing base to reduce glycolytic metabolism and viability of de novo plaque bacteria using the plaque glycolysis regrowth model (PGRM).

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon oral examination.
* Plaque sample acidogenicity in the pH range 5.0 to 5.7 at Visit.

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding.
* Currently taking antibiotics or have taken antibiotics within 2 weeks of plaque assessment (Visit 2). A participant with any medical history that may prevent them from participating in the study until study conclusion (such as diabetes).
* Any sign of grossly carious lesions (active), moderate or severe periodontal conditions, or severe tooth wear.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Current smokers, or smokers who have quit within 6 months of screening, or participants currently using smokeless forms of tobacco, e.g. Gutkha, Pan containing tobacco, Pan Masala.
* Current active caries or periodontitis that may compromise, in the opinion of the investigator, study outcomes or the health of the subject.
* Restorations in a poor state of repair that may, in the opinion of the investigator, compromise study outcomes or the health of the participant.
* Partial dentures or orthodontic appliances that may, in the opinion of the investigator, compromise study outcomes or the health of the participant.
* Recent history (within the last year) of alcohol or other substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 150 participants were screened, of which 45 participants were randomized and 44 completed the study.
Groups:
- Overall Study: This was a single-centre, analyst and examiner (plaque sample collector)-blind, randomized, five-treatment, five-period, cross-over study in healthy adult participants. Each participant received each of the five interventions i.e., Test Zinc-isopropylmethylphenol (IPMP), Test Zinc non-IPMP, Positive control, non-sodium lauryl sulphate (SLS) negative control, SLS negative control.
Period: Overall Study
Arm/Group | Overall Study
Started | 45
Received Test Zinc-IPMP | 44
Received Test Zinc Non-IPMP | 44
Received Positive Control | 45
Received Non-SLS Negative Control | 44
Received SLS Negative Control | 44
Completed | 44
Not Completed | 1
Not completed — Withdrawal of consent | 1

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were included for baseline evaluation.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.4 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve for Glycolysis (AUCgly(0-90)) of Test Zinc-IPMP and Non-SLS Negative Control
Description: AUCgly(0-90) of Test zinc-IPMP and non-SLS negative control was calculated using trapezoidal method.
Time Frame: Baseline up to 90 minutes (min)
Population: The Per Protocol (PP) population defined as those participants in the intent to treat (ITT) population who had at least one assessment of efficacy considered unaffected by protocol violation.
Measure: Least Squares Mean (Standard Error); unit: plaque incubation pH*min
Groups:
- Test Zinc-IPMP: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 0.454% w/w stannous fluoride (1100 ppm F as stannous fluoride) in 10 mL water for 60 sec followed by rinse with 10 mL water
- Non-SLS Negative Control: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 1426 ppm F as sodium fluoride in 10 mL water for 60 sec followed by rinse with 10 mL water
Arm/Group | Test Zinc-IPMP | Non-SLS Negative Control
Number analyzed (Participants) | 14 | 15
plaque incubation pH*min | 42.64 (3.437) | 2.46 (3.303)
Statistical Analysis 1: Comparison: Test Zinc-IPMP vs Non-SLS Negative Control; Test type: Superiority or Other; p < 0.0001, ANCOVA — Obtained from ANCOVA including period and treatment as fixed effects, participant as a random effect and participant-level pre-treatment values and period minus participant-level pre-treatment values as covariates in the model; Least square (LS) mean difference = 40.18, 95% CI 2-sided [32.37 to 47.99] — Difference is first named treatment minus second named treatment such that a positive difference indicates a greater inhibition of plaque Glycolysis for the first named treatment

2. Secondary Outcome: AUCgly(0-90) for Test Zinc-IPMP, Test Zinc Non-IPMP, Positive Control, Non-SLS Negative Control and SLS Negative Control
Description: AUCgly(0-90) for test zinc-IPMP, test zinc non-IPMP, positive control, non-SLS negative control and SLS negative control was calculated using trapezoidal method.
Time Frame: Baseline up to 90 min
Population: PP population defined as those participants in the ITT population who had at least one assessment of efficacy considered unaffected by protocol violation.
Measure: Least Squares Mean (Standard Error); unit: plaque incubation pH*min
Groups:
- Test Zinc-IPMP: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 0.6% w/w zinc chloride and 0.1% w/w IPMP and 1426ppm F as sodium fluoride in 10mL water for 60 sec followed by rinse with 10mL water
- Test Zinc Non- IPMP: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 0.6% w/w zinc chloride and 0% w/w IPMP and 1426ppm F as sodium fluoride in 10mL water for 60 sec followed by rinse with 10mL water
- Positive Control: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 0.454% w/w stannous fluoride (1100ppm F as stannous fluoride) in 10mL water for 60 sec followed by rinse with 10mL water
- Non-SLS Negative Control: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 1426ppm F as sodium fluoride in 10mL water for 60 sec followed by rinse with 10mL water
- SLS Negative Control: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 2.0% SLS, 0.65% Tegobetain and 1150ppm fluoride as sodium fluoride in 10mL water for 60 sec followed by rinse with 10mL water
Arm/Group | Test Zinc-IPMP | Test Zinc Non- IPMP | Positive Control | Non-SLS Negative Control | SLS Negative Control
Number analyzed (Participants) | 14 | 14 | 14 | 15 | 14
plaque incubation pH*min | 42.64 (3.437) | 34.20 (3.354) | 28.88 (3.384) | 2.46 (3.303) | 31.78 (3.512)
Statistical Analysis 1: Comparison: Positive Control vs Non-SLS Negative Control; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 26.41, 95% CI 2-sided [18.94 to 33.88] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Positive Control vs SLS Negative Control; Test type: Superiority or Other; p = 0.4823, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -2.91, 95% CI 2-sided [-11.18 to 5.37] — Difference is first named treatment minus second named treatment such that a positive difference indicates a greater inhibition of glycolysis for the first named treatment
Statistical Analysis 3: Comparison: Test Zinc-IPMP vs SLS Negative Control; Test type: Superiority or Other; p = 0.0072, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 10.86, 95% CI 2-sided [3.13 to 18.59] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Test Zinc-IPMP vs Positive Control; Test type: Superiority or Other; p = 0.0009, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 13.77, 95% CI 2-sided [6.01 to 21.53] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Test Zinc-IPMP vs Test Zinc Non- IPMP; Test type: Superiority or Other; p = 0.0286, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 8.44, 95% CI 2-sided [0.93 to 15.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Test Zinc Non- IPMP vs Positive Control; Test type: Superiority or Other; p = 0.1573, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 5.32, 95% CI 2-sided [-2.15 to 12.79] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Non-SLS Negative Control vs SLS Negative Control; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -29.32, 95% CI 2-sided [-37.20 to -21.43] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Test Zinc Non- IPMP vs Non-SLS Negative Control; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 31.74, 95.0% CI 2-sided [24.18 to 39.30] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Test Zinc Non- IPMP vs SLS Negative Control; Test type: Superiority or Other; p = 0.5174, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 2.42, 95% CI 2-sided [-5.08 to 9.92] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: AUCregrowth(0-90) for Test Zinc-IPMP, Test Zinc Non-IPMP, Positive Control, Non-SLS Negative Control and SLS Negative Control
Description: AUCregrowth(0-90) for test zinc-IPMP, test zinc non-IPMP, positive control, non-SLS negative control and SLS negative control was calculated using trapezoidal method.
Time Frame: Baseline up to 90 min
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: regrowth ratio*min
Arm/Group | Test Zinc-IPMP | Test Zinc Non- IPMP | Positive Control | Non-SLS Negative Control | SLS Negative Control
Number analyzed (Participants) | 14 | 14 | 14 | 15 | 14
regrowth ratio*min | -239.81 (40.122) | -240.86 (39.118) | -179.55 (39.415) | 53.66 (38.443) | -215.08 (40.350)
Statistical Analysis 1: Comparison: Positive Control vs Non-SLS Negative Control; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -233.22, 95% CI 2-sided [-332.88 to -133.55] — Difference is first named treatment minus second named treatment such that a negative difference indicates a greater inhibition of plaque regrowth for the first named treatment
Statistical Analysis 2: Comparison: Positive Control vs SLS Negative Control; Test type: Superiority or Other; p = 0.5018, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 35.53, 95% CI 2-sided [-69.90 to 140.96] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Test Zinc-IPMP vs SLS Negative Control; Test type: Superiority or Other; p = 0.6325, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -24.73, 95% CI 2-sided [-128.07 to 78.61] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Test Zinc-IPMP vs Positive Control; Test type: Superiority or Other; p = 0.2427, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -60.26, 95% CI 2-sided [-162.72 to 42.21] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Test Zinc-IPMP vs Test Zinc Non- IPMP; Test type: Superiority or Other; p = 0.9834, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 1.05, 95% CI 2-sided [-100.50 to 102.61] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Test Zinc Non- IPMP vs Positive Control; Test type: Superiority or Other; p = 0.2226, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -61.31, 95% CI 2-sided [-161.14 to 38.52] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Non-SLS Negative Control vs SLS Negative Control; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 268.74, 95% CI 2-sided [165.98 to 371.51] — Difference is second named treatment(non-SLS negative control) minus first named treatment (SLS negative control) such that a negative difference indicates a greater inhibition of plaque
Statistical Analysis 8: Comparison: Test Zinc-IPMP vs Non-SLS Negative Control; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -293.47, 95% CI 2-sided [-396.03 to -190.91] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Test Zinc Non- IPMP vs Non-SLS Negative Control; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -294.53, 95% CI 2-sided [-395.43 to -193.62] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: Test Zinc Non- IPMP vs SLS Negative Control; Test type: Superiority or Other; p = 0.6086, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -25.78, 95% CI 2-sided [-126.53 to 74.96] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: AUClive:Dead(0-90) for Test Zinc-IPMP, Test Zinc Non-IPMP, Positive Control, Non-SLS Negative Control and SLS Negative Control
Description: AUClive:dead(0-90) for test zinc-IPMP, test zinc non-IPMP, positive control, non-SLS negative control and SLS negative control was calculated using trapezoidal method.
Time Frame: Baseline up to 90 min
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: live:dead stain ratio*min
Groups:
- Test Zinc-IPMP: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 0.6% w/w zinc chloride and 0.1% w/w IPMP and 1426 ppm F as sodium fluoride in 10 mL water for 60 sec followed by rinse with 10 mL water
- Test Zinc Non- IPMP: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 0.6% w/w zinc chloride and 0% w/w IPMP and 1426 ppm F as sodium fluoride in 10 mL water for 60 sec followed by rinse with 10 mL water
- Positive Control: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 0.454% w/w stannous fluoride (1100 ppm F as stannous fluoride) in 10 mL water for 60 sec followed by rinse with 10 mL water
- SLS Negative Control: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 2.0% SLS, 0.65% Tegobetain and 1150 ppm fluoride as sodium fluoride in 10 mL water for 60 sec followed by rinse with 10 mL water
Arm/Group | Test Zinc-IPMP | Test Zinc Non- IPMP | Positive Control | Non-SLS Negative Control | SLS Negative Control
Number analyzed (Participants) | 9 | 10 | 11 | 14 | 12
live:dead stain ratio*min | 75.23 (568.834) | -691.41 (508.108) | 72.19 (491.718) | 346.11 (431.974) | -601.87 (499.740)
Statistical Analysis 1: Comparison: Positive Control vs Non-SLS Negative Control; Test type: Superiority or Other; p = 0.6664, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -273.92, 95% CI 2-sided [-1550.45 to 1002.61] — Difference is first named treatment minus second named treatment such that a negative difference indicates a smaller live:dead stain ratio for the first named treatment
Statistical Analysis 2: Comparison: Positive Control vs SLS Negative Control; Test type: Superiority or Other; p = 0.3249, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 674.06, 95% CI 2-sided [-692.21 to 2040.33] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Test Zinc-IPMP vs SLS Negative Control; Test type: Superiority or Other; p = 0.3544, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 677.09, 95% CI 2-sided [-784.16 to 2138.35] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Test Zinc-IPMP vs Positive Control; Test type: Superiority or Other; p = 0.9967, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 3.04, 95% CI 2-sided [-1469.45 to 1475.52] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Test Zinc-IPMP vs Test Zinc Non- IPMP; Test type: Superiority or Other; p = 0.2976, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 766.64, 95% CI 2-sided [-703.26 to 2236.54] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Test Zinc Non- IPMP vs Positive Control; Test type: Superiority or Other; p = 0.2702, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -763.60, 95% CI 2-sided [-2144.45 to 617.25] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Non-SLS Negative Control vs SLS Negative Control; Test type: Superiority or Other; p = 0.1511, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 947.97, 95% CI 2-sided [-361.95 to 2257.90] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Test Zinc-IPMP vs Non-SLS Negative Control; Test type: Superiority or Other; p = 0.6998, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -270.88, 95% CI 2-sided [-1680.58 to 1138.82] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Test Zinc Non- IPMP vs Non-SLS Negative Control; Test type: Superiority or Other; p = 0.1210, ANCOVA — Obtained from ANCOVA including period and treatment as fixed effects, participant as a random effect and participant -level pre-treatment values and period minus participant -level pre-treatment values as covariates in the model; LS mean difference = -1037.52, 95% CI 2-sided [-2361.33 to 286.29] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: Test Zinc Non- IPMP vs SLS Negative Control; Test type: Superiority or Other; p = 0.8935, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -89.54, 95% CI 2-sided [-1439.50 to 1260.41] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Groups:
- Test Zinc-IPMP Toothpaste: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 0.6% w/w zinc chloride and 0.1% w/w IPMP and 1426 ppm F as sodium fluoride in 10 mL water for 60 sec followed by rinse with 10 mL water
- Test Zinc Non- IPMP Toothpaste: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 0.6% w/w zinc chloride and 0% w/w IPMP and 1426 ppm F as sodium fluoride in 10 mL water for 60 sec followed by rinse with 10 mL water
- Positive Control Toothpaste: Participants were instructed to rinse their mouth with prepared slurry of toothpaste containing 0.454% w/w stannous fluoride (1100 ppm F as stannous fluoride) in 10 mL water for 60 sec followed by rinse with 10 mL water
Arm/Group | Test Zinc-IPMP Toothpaste | Test Zinc Non- IPMP Toothpaste | Positive Control Toothpaste | Non-SLS Negative Control | SLS Negative Control
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44 | 0/45 | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 8/44 | 6/44 | 6/45 | 3/44 | 2/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Zinc-IPMP Toothpaste (N=44) | Test Zinc Non- IPMP Toothpaste (N=44) | Positive Control Toothpaste (N=45) | Non-SLS Negative Control (N=44) | SLS Negative Control (N=44)
LIP ULCERATION (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
PARAESTHESIA ORAL (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
TOOTHACHE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
COATING IN MOUTH (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
GINGIVAL ULCERATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
RHINITIS (Infections and infestations) | 1 | 1 | 2 | 2 | 1
ORAL HERPES (Infections and infestations) | 0 | 1 | 0 | 0 | 0
PERICORONITIS (Infections and infestations) | 0 | 1 | 1 | 0 | 0
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
SUPERFICIAL INJURY OF EYE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
DEVICE FAILURE (General disorders) | 0 | 0 | 0 | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.